CLINICAL TRIAL: NCT00053027
Title: Phase II Trial of Rituximab and 2-Chlorodeoxyadenosine (2-CDA) in Newly Diagnosed Mantle Cell Lymphoma (MCL)
Brief Title: Rituximab and Cladribine in Treating Patients With Newly Diagnosed Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-N0189; NCI-2012-02510 (Registry Identifier: NCI-2012-02510 CTRP (Clinical Trials Reporting System)); CDR0000269055 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2003-01-27; First posted 2003-01-28 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-12

CONDITIONS: Lymphoma
Keywords: contiguous stage II mantle cell lymphoma; noncontiguous stage II mantle cell lymphoma; stage I mantle cell lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Mantle-Cell | interventions — Rituximab; Cladribine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- rituximab + cladribine (Experimental): Patients receive rituximab IV over 4-8 hours on day 1 and cladribine IV over 2 hours on days 4-8. If 2 or more patients experience unacceptable toxicity during the first course, the study is discontinued; otherwise, the study is opened for enrollment at all NCCTG sites.
  Treatment repeats every 28 days for a total of 2-6 courses in the absence of disease progression or unacceptable toxicity.
  Patients are followed every 2 months for 1 year, every 4 months for 1 year, every 6 months for 1 year, and then annually for 2 years.
  Interventions: Biological: rituximab; Drug: cladribine

INTERVENTIONS:
Biological: rituximab
Drug: cladribine

SUMMARY:
RATIONALE: Monoclonal antibodies such as rituximab can locate cancer cells and either kill them or deliver cancer-killing substances to them without harming normal cells. Drugs used in chemotherapy such as cladribine work in different ways to stop cancer cells from dividing so they stop growing or die. Combining rituximab with cladribine may kill more cancer cells.

PURPOSE: This phase II trial is studying how well giving rituximab together with cladribine works in treating patients with newly-diagnosed mantle cell lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether rituximab and cladribine will increase the complete remission rate and the unconfirmed complete remission rate in patients with mantle cell lymphoma.
* Determine the time to progression in patients treated with this regimen.
* Determine the toxic effects of this regimen in these patients.

OUTLINE: This is a multicenter study.

An initial cohort of 6 patients at Mayo Clinic receives rituximab IV over 4-8 hours on day 1 and cladribine IV over 2 hours on days 4-8. If 2 or more patients experience unacceptable toxicity during the first course, the study is discontinued; otherwise, the study is opened for enrollment at all NCCTG sites. (The phase II study is open for enrollment as of 5/14/04.)

Treatment repeats every 28 days for a total of 2-6 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed every 2 months for 1 year, every 4 months for 1 year, every 6 months for 1 year, and then annually for 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed mantle cell lymphoma*
* Measurable or assessable disease defined as at least one of the following:

  * Lymph node or tumor mass that is 2.0 cm or more in at least one dimension by CT scan, MRI, or plain radiograph imaging OR greater than 1.5 cm in at least one dimension by physical exam
  * Splenic enlargement, if the spleen is palpable, at least 3 cm below the left costal margin
  * Diffuse infiltration of an organ such as the stomach, bone marrow, peripheral blood, liver, lungs, or bowel by lymphoma without a discrete mass would constitute assessable, but not measurable, disease
* No known CNS involvement NOTE: *If tumor tissue is unavailable for biopsy, blood or bone marrow specimens may be used to establish patient eligibility provided fusion signals indicate the presence of t(11;14)(q13;q32) by fluorescence in situ hybridization using CCND1/IGH AND mantle cell lymphoma involvement is determined by morphology

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-3

Life expectancy

* At least 12 weeks

Hematopoietic

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic

* Total or direct bilirubin no greater than upper limit of normal (ULN) (with or without secondary liver involvement)
* SGOT no greater than 3 times ULN (5 times ULN if there is liver involvement)

Renal

* Creatinine no greater than 2.0 mg/dL

Cardiovascular

* No myocardial infarction within the past 6 months
* No uncontrolled high blood pressure
* No unstable angina
* No serious uncontrolled cardiac arrhythmia
* No active congestive heart failure

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 30 days after study participation
* HIV negative
* No other malignancy within the past 5 years except carcinoma in situ of the cervix, resected basal cell or squamous cell skin cancer, or prostate cancer that is in remission after a radical retropubic prostatectomy or radiotherapy
* No medical or psychiatric condition that makes the patient a poor risk for this study
* No active or uncontrolled infection
* No known hypersensitivity to rituximab or its components or to murine proteins

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior biologic therapy for mantle cell lymphoma

Chemotherapy

* No prior chemotherapy for mantle cell lymphoma

Endocrine therapy

* No prior endocrine therapy for mantle cell lymphoma

Radiotherapy

* No prior radiotherapy

Surgery

* Prior splenectomy allowed (for diagnosis, cytopenia, or symptomatic splenomegaly)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2003-02; Primary Completion 2006-01 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Complete remission (CR) and complete remission unconfirmed (CRu) rate at the close of study therapy assessment (after 2, 4, or 6 courses) | Up to 4 years

SECONDARY OUTCOMES:
Progression at any time after therapy | Up to 4 years

CONTACTS AND LOCATIONS:
Overall Officials: David J. Inwards, MD, Study Chair — Mayo Clinic

REFERENCES:
- [Background] Inwards DJ, Fishkin PA, Hillman DW, Brown DW, Ansell SM, Kurtin PJ, Fonseca R, Morton RF, Veeder MH, Witzig TE. Long-term results of the treatment of patients with mantle cell lymphoma with cladribine (2-CDA) alone (95-80-53) or 2-CDA and rituximab (N0189) in the North Central Cancer Treatment Group. Cancer. 2008 Jul 1;113(1):108-16. doi: 10.1002/cncr.23537. PMID 18470909